CLINICAL TRIAL: NCT06974851
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled Clinical Study to Evaluate the Efficacy and Safety of HRS9531 Injection in Subjects With Obstructive Sleep Apnea (OSA) and Obesity Not Receiving Positive Airway Pressure (PAP) Therapy
Brief Title: A Phase III Study Evaluating the Efficacy and Safety of HRS9531 Injection in Subjects With Obstructive Sleep Apnea (OSA) and Obesity
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS9531-306
Record Dates: First submitted 2025-04-24; First posted 2025-05-16 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-04

CONDITIONS: Bstructive Sleep Apnea (OSA) and Obesity
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: HRS9531 (Experimental)
  Interventions: Drug: HRS9531
- Group 2: HRS9531placebo (Placebo Comparator)
  Interventions: Drug: HRS9531placebo

INTERVENTIONS:
Drug: HRS9531 — HRS9531
  Arms: Group 1: HRS9531
Drug: HRS9531placebo — HRS9531placebo
  Arms: Group 2: HRS9531placebo

SUMMARY:
A Phase III Study Evaluating the Efficacy and Safety of HRS9531 Injection in Subjects with Obstructive Sleep Apnea (OSA) and Obesity

ELIGIBILITY:
Inclusion Criteria:

1. The participant has provided informed consent and is willing and able to comply with the study protocol requirements to complete the study.
2. Age between 18 and 75 years, male or female, at the time of signing the informed consent form.
3. BMI ≥ 28.0 kg/m² at screening.
4. Has been on a controlled diet and exercise regimen for 3 months or more, with a weight change of ≤ 5.0 kg in the past 3 months.
5. Polysomnography (PSG) results at screening confirm OSA.
6. Female participants of childbearing potential and male participants with partners of childbearing potential agree to use highly effective contraception from the time of signing the informed consent form until 2 months after the last dose, with no plans for pregnancy or donation of eggs/sperm during this period. Female participants of childbearing potential must have a negative pregnancy test within 3 days prior to randomization and must not be breastfeeding.

Exclusion Criteria:

1. Laboratory Test Abnormalities:

   1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 3 × upper limit of normal (ULN), or total bilirubin (TBIL) ≥ 2.0 × ULN.
   2. Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m² (calculated using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula based on serum creatinine).
   3. Thyroid-stimulating hormone (TSH) < 0.4 or > 6.0 mIU/L.
   4. Other laboratory abnormalities judged by the investigator to potentially affect efficacy or safety assessments.
2. Clinically Significant ECG Abnormalities:

   ECG findings deemed clinically significant by the investigator, including but not limited to myocardial infarction, severe arrhythmias (e.g., supraventricular tachycardia, atrial fibrillation, atrial flutter, second- or third-degree atrioventricular block, etc.), which may affect participant safety.
3. Poorly Controlled Blood Pressure:

   Systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg.
4. PHQ-9 Score ≥ 15:

   Patient Health Questionnaire-9 (PHQ-9) score ≥ 15.
5. Medical History or Conditions Prior to Screening or Randomization:

   1. Endocrine disorders or monogenic mutations causing obesity or hereditary obesity syndromes that may significantly affect weight.
   2. Diabetes mellitus.
   3. Diagnosis of central or mixed sleep apnea or Cheyne-Stokes respiration.
   4. Respiratory or neuromuscular diseases judged by the investigator to potentially interfere with trial results.
   5. Clinical abnormalities or diseases related to insomnia or excessive sleepiness (excluding OSA).
   6. History of conditions affecting gastric emptying, long-term use of medications directly affecting gastrointestinal motility, severe gastrointestinal diseases, or prior gastrointestinal surgery.
   7. History of acute or chronic pancreatitis, pancreatic injury, acute cholecystitis, or symptomatic/treatment-requiring gallbladder disease.
   8. Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN2).
   9. Severe infections, significant trauma, or major/moderate surgery within 1 month prior to screening.
   10. Severe cardiovascular or cerebrovascular events within 6 months prior to screening, including decompensated heart failure (NYHA Class III or IV), unstable angina, stroke or transient ischemic attack, myocardial infarction, severe arrhythmias, or cardiac surgeries such as coronary artery bypass grafting or percutaneous coronary intervention.
   11. Malignancy in any organ system within the past 5 years, regardless of evidence of local recurrence or metastasis (except cured local basal cell carcinoma, cervical carcinoma in situ, and prostate carcinoma in situ).
   12. Presence or suspicion of depression, bipolar disorder, suicidal tendencies, schizophrenia, or other severe psychiatric disorders.
   13. Known or suspected history of alcohol and/or drug abuse or drug addiction.
   14. Acute or chronic hepatitis or other severe liver diseases (excluding non-alcoholic fatty liver disease).
   15. Severe hematologic diseases (e.g., aplastic anemia, myelodysplastic syndrome, hemolytic anemia, sickle cell disease) or any condition causing hemolysis or red blood cell instability (e.g., malaria).
   16. Autoimmune diseases requiring systemic corticosteroid or immunosuppressive therapy during the study period.
6. Medications or Treatments Prior to Screening:

   1. Use of medications or treatments likely to cause significant weight gain or loss within 3 months prior to screening.
   2. Medications or treatments judged by the investigator to potentially affect sleepiness assessments.
   3. Prior or planned bariatric surgery (except liposuction performed more than 1 year ago).
   4. Prior or planned endoscopic or device-based weight loss treatments, or device removal within the past 6 months (e.g., mucosal ablation, gastric artery embolization, intragastric balloons, duodenal-jejunal bypass sleeves).
   5. Use of positive airway pressure (PAP) or other OSA treatments judged by the investigator to potentially interfere with study results (e.g., oral appliances, neurostimulation therapy), unless the participant is willing to discontinue such treatments 4 weeks prior to screening and during the study.
   6. Requirement for supplemental oxygen.
7. Other Exclusion Criteria:

   1. Participation in any drug or medical device clinical trial within 3 months prior to screening, defined as signing informed consent and using the investigational product (including placebo) or medical device, or still within 5 half-lives of the investigational drug (whichever is longer).
   2. History of blood donation or blood loss ≥ 400 mL within 3 months prior to screening, or receipt of a blood transfusion within 3 months.
   3. Planned surgery during the trial (except minor surgeries deemed by the investigator to not affect the trial).
   4. Participants with mental incapacity or language barriers unable to fully understand or participate in the trial.
   5. Any condition judged by the investigator to affect participant safety or interfere with the evaluation of trial results (medical, psychological, social, or geographical factors, etc.).
   6. Investigators, research site staff, or other individuals directly involved in the execution of the protocol, and their immediate family members (e.g., spouse, legal partner, parents, children, or siblings). Employees of Hengrui Company are also excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage Change in AHI from Baseline at Week 52 of Treatment | 52week

SECONDARY OUTCOMES:
Changes in AHI Relative to Baseline After 52 Weeks of Treatment | 52week
Proportion of Subjects with AHI <5.0 events/h, or AHI 5.0-14.0 events/h with Epworth Sleepiness Scale (ESS) ≤10 at Week 52 of Treatment | 52week
Percentage Change in Body Weight from Baseline at Week 52 of Treatment | 52week
Change in Epworth Sleepiness Scale (ESS) Score from Baseline at Week 52 of Treatment | 52week
Proportion of Subjects Achieving ≥5%, ≥10%, ≥15%, and ≥20% Reduction in Body Weight from Baseline at Week 52 of Treatment | 52week
Change in Body Weight and Body Mass Index (BMI) from Baseline at Week 52 of Treatment | 52week
Change in systolic and diastolic blood pressure from baseline at Week 52 of treatment. | 52week
Proportion of subjects reporting improvement in Patient Global Impression of Severity (PGIS)-OSA categories (sleepiness, fatigue, snoring) at Week 52 of treatment. | 52week
Incidence of adverse events (AEs) | 52week

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided